CLINICAL TRIAL: NCT06794905
Title: Comparing Hartmann's Procedure and Primary Resection with Anastomosis in Hinchey III-IV Diverticulitis: Focus on Ostomy Closure and Long-Term Outcomes
Acronym: ARES
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, Principal Investigator, PhD, Md, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 20252818
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Diverticular Disease of Colon; Colostomy Complication; Colostomy - Stoma
Keywords: Hartmann; Diverticular Disease of colon; stoma
MeSH Terms: conditions — Diverticulosis, Colonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- rimary Anastomosis with Diverting Loop Ileostomy Group: This group includes patients who underwent segmental resection of the sigmoid colon followed by primary end-to-end anastomosis, protected by a diverting loop ileostomy. The surgical approach aimed to restore bowel continuity while minimizing the risk of anastomotic leakage through the protective ileostomy. Patients in this group were typically stable at the time of surgery, with no life-threatening sepsis or severe hemodynamic instability. Key metrics evaluated included stoma reversal rates, time to stoma closure, postoperative complications (both surgical and systemic), length of hospital stay, and quality of life after recovery. The technical approach incorporated the double-stapling method for anastomosis, and structured follow-up was implemented to monitor for dehydration, electrolyte imbalances, and long-term outcomes such as hernias and recurrence.
- Hartmann's Procedure Group: This group comprises patients who underwent segmental resection of the sigmoid colon with the creation of an end colostomy, leaving the distal rectal stump closed. Hartmann's procedure was performed primarily in patients with more severe clinical conditions, including those with significant sepsis or hemodynamic instability, where the risk of anastomotic complications was deemed unacceptably high. Outcomes assessed in this group included the rates of permanent colostomy, incidence of parastomal hernias, long-term complications related to the colostomy, and overall recovery metrics. Patients were evaluated for potential stoma reversal, although a significant proportion of individuals in this group retained a permanent stoma due to either clinical contraindications or patient preference. Structured follow-up focused on addressing colostomy-related challenges and minimizing complications.

SUMMARY:
Brief Summary

This multicenter study compares the effectiveness of primary anastomosis with diverting loop ileostomy to Hartmann's procedure for managing perforated sigmoid diverticulitis in stable patients. The findings demonstrate that primary anastomosis with diverting loop ileostomy offers superior long-term outcomes, including higher stoma reversal rates (92% versus 58%), shorter time to closure, and fewer parastomal hernias, contributing to improved quality of life. Kaplan-Meier analysis further supports the benefits of primary anastomosis with diverting loop ileostomy, showing significantly better stoma-free survival rates at 24 months. Despite higher short-term readmission rates due to ileostomy-related complications, patients undergoing primary anastomosis with diverting loop ileostomy experienced shorter hospital stays and fewer long-term complications compared to patients undergoing Hartmann's procedure. While Hartmann's procedure remains crucial for unstable cases, the functional and psychological advantages of primary anastomosis with diverting loop ileostomy underscore its value for stable patients. Future research should focus on randomized trials and minimally invasive approaches to refine surgical strategies.

DETAILED DESCRIPTION:
Detailed Description

This multicenter study evaluates and compares the outcomes of primary anastomosis with diverting loop ileostomy and Hartmann's procedure in the surgical management of perforated sigmoid diverticulitis in stable patients. Conducted across multiple surgical centers, the study provides a comprehensive overview of these approaches in real-world clinical settings. The findings indicate that primary anastomosis with diverting loop ileostomy demonstrates significant advantages over Hartmann's procedure, particularly in terms of long-term outcomes, stoma management, and recovery metrics.

Patients who underwent primary anastomosis with diverting loop ileostomy achieved notably higher stoma reversal rates (92% versus 58%), a shorter median time to stoma closure, and fewer stoma-related complications such as parastomal hernias. These results underscore the benefits of restoring bowel continuity, which plays a critical role in improving both physical functionality and psychological well-being. Kaplan-Meier analysis confirmed superior stoma-free survival rates at 24 months for patients receiving primary anastomosis with diverting loop ileostomy compared to those treated with Hartmann's procedure.

While Hartmann's procedure remains a valuable option for unstable or critically ill patients due to its simplicity, its long-term disadvantages include a higher prevalence of stoma-related complications, such as parastomal hernias and challenges with colostomy management. Conversely, primary anastomosis with diverting loop ileostomy was associated with a slightly higher rate of early readmissions, often due to issues related to the protective ileostomy, including dehydration and electrolyte imbalances. However, these complications were generally manageable with appropriate follow-up care.

The study also highlights shorter hospital stays and faster recovery times for patients treated with primary anastomosis with diverting loop ileostomy, contributing to reduced healthcare costs and improved quality of life. These findings suggest that primary anastomosis with diverting loop ileostomy should be considered a first-line option for stable patients, with Hartmann's procedure reserved for those in critical conditions. Future research is recommended to further investigate minimally invasive techniques, long-term quality of life outcomes, and randomized controlled trials to solidify these findings and refine surgical practices.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosed with perforated sigmoid diverticulitis classified as Hinchey Stage III or IV.
* Clinically stable patients suitable for emergency colonic resection.
* Eligible to undergo either primary anastomosis with diverting loop ileostomy or Hartmann's procedure.
* Provided informed consent or had a legal surrogate able to consent on their behalf.

Exclusion Criteria:

* Hinchey Stage I or II diverticulitis, typically managed conservatively or with less invasive interventions.
* Postoperative confirmation of malignancy as the primary cause of the perforation.
* Undergoing laparoscopic surgery rather than open resection.
* Clinically unstable patients with severe sepsis, septic shock, or significant hemodynamic compromise.
* Pre-existing stomas or prior colonic resections.
* Significant comorbidities, such as advanced cardiac or respiratory failure.
* Limited life expectancy due to terminal illnesses (e.g., advanced malignancies).
* Inability to participate in follow-up assessments due to cognitive impairments or logistical barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults presenting with acute perforated sigmoid diverticulitis at five surgical centers across Italy, encompassing both academic and community hospitals. This population represents a diverse cohort of patients encountered in real-world clinical settings, allowing for a broad evaluation of outcomes across varying levels of healthcare infrastructure and expertise.
  Participants will be selected from patients admitted through emergency departments with a confirmed diagnosis of perforated sigmoid diverticulitis classified as Hinchey Stage III or IV. The population includes clinically stable individuals who are eligible for emergency surgical intervention and capable of undergoing either primary anastomosis with diverting loop ileostomy or Hartmann's procedure. The inclusion of patients from different regions and centers ensures a heterogeneous sample that reflects diverse demographic, socioeconomic, and clinical characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Stoma closure within 24 months | 24 months
  This outcome was chosen for its significant impact on patient quality of life and its role in reflecting the resolution of temporary stomas created during the initial surgery. Achieving stoma closure minimizes long-term stoma-related complications such as parastomal hernias, psychosocial distress, and reduced functionality. The study evaluates not only whether stoma closure occurs but also the time to closure, perioperative complications, and factors influencing closure feasibility, offering a comprehensive view of patient recovery.

SECONDARY OUTCOMES:
Surgical Complications | 24 months
  Surgery-specific complications: Rates of anastomotic leaks, intra-abdominal abscesses, surgical site infections, delayed healing, and hemorrhage.
Index Admission Outcomes | 24 months
  Length of hospital stay, stratified by procedure type.

IPD SHARING:
Plan to Share IPD: Undecided
The study will include all de-identified individual participant data (IPD) supporting the results, such as demographic, clinical, surgical, and follow-up information, including quality of life and long-term follow-up data. A decision on IPD sharing is pending, considering patient privacy, data ownership, and compliance with GDPR and ethical regulations. Data sharing may be possible upon reasonable request to qualified researchers through secure agreements after further evaluation.

REFERENCES:
- [Background] Rehmani S, Bhora F, Flores R. Robotic Lung Cancer Surgery: A Missed Opportunity and a Faulty Conclusion. Ann Surg. 2018 Feb;267(2):e34. doi: 10.1097/SLA.0000000000001996. No abstract available. PMID 27643927